CLINICAL TRIAL: NCT05247437
Title: A Pilot Cluster Randomized Controlled Trial of a Digital Lifestyle Intervention for Individuals With Prediabetes or Type 2 Diabetes
Brief Title: Digital Lifestyle Intervention For Diabetes/Pre-Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Wai Sze, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA220053
Record Dates: First submitted 2022-01-28; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes; PreDiabetes; Obesity
Keywords: Intensive Lifestyle Intervention; mHealth; eHealth; digital intervention; efficacy; RCT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Obesity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FitD full version (Experimental)
  Interventions: Behavioral: Digital Intensive Lifestyle Intervention
- Digital Self-Help (Active Comparator)
  Interventions: Behavioral: Digital Self-Help Control Condition

INTERVENTIONS:
Behavioral: Digital Intensive Lifestyle Intervention — The FitD consists of 8 digital lessons on how to improve dietary and exercise habits using self-monitoring, goal-setting, cognitive restructuring, and other behavioral and cognitive strategies. The FitD app offers a virtual coach that guides the participant to complete the treatment.
  Arms: FitD full version
Behavioral: Digital Self-Help Control Condition — The digital self-help control condition consists of educational materials related to diet and exercise. The materials are open for access all at once. There is no guidance by a virtual coach or digital lessons.
  Arms: Digital Self-Help

SUMMARY:
The study aims to evaluate the acceptability, feasibility, and preliminary efficacy of a digital lifestyle intervention, called Fitness Digital (FitD), for individuals with prediabetes or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Hong Kong resident
* Can understand Chinese and Cantonese
* Have self-reported diagnosis of type 2 diabetes or prediabetes
* Have a smart phone and able to use a mobile app

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-19 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the scores on the Summary of Diabetes Self-Care Activities - Revised (SDSCA) | Baseline (week 0), posttreatment (week 9), follow-up (week 21)
  The Summary of Diabetes Self-Care Activities consists of 11 items asking the frequency of diabetes self-care behavior in the following six areas: general diet, specific diet (ate fruit and vegetable/ low fat diet), exercise, blood glucose testing, foot care, and cigarette smoking. The maximum score is 70 and the minimum score is 0. A higher total score indicate better self-care.
Changes in weight from baseline (week 0) to posttreatment (week 9) | Baseline (week 0), posttreatment (week 9), follow-up (week 21)
  Self-reported weight in kilograms

SECONDARY OUTCOMES:
Changes in the scores on the Weight Control Strategy Scale | Baseline (week 0), posttreatment (week 9), follow-up (week 21)
  The Weight Control Strategy Scale consists of 30 items measuring one's use of different weight control strategies. A higher score indicates greater use of effective weight control strategies.
Changes in the scores on the Physical activity acceptance and action questionnaire | Baseline (week 0), posttreatment (week 9), follow-up (week 21)
  The Physical activity acceptance and action questionnaire consists of 10 items assessing one's readiness and motivation to engage in increased physical activity. A higher score indicates greater readiness and motivation.
Changes in the scores on the Weight loss self-efficacy scale | Baseline (week 0), posttreatment (week 9), follow-up (week 21)
  The weight loss self-efficacy scale consists of 10 items assessing one's confidence in using effective strategies for weight loss. A higher score indicates greater confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Sze Chan, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available for sharing upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: During review of or after the publication of the study findings.
Access Criteria: For other research teams' secondary analysis